CLINICAL TRIAL: NCT07019350
Title: Drug-Coated Balloon Versus Drug-eluting Stent for Treatment of Clinically Relevant Side Branch in Complex Coronary Bifurcation Lesion
Brief Title: Smart Angioplasty Research Team-Optimal Strategy for Side Branch Stenting in Coronary Bifurcation Lesion With Drug-Coated Balloon
Acronym: SMART-DCB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Bin Song, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMC-SMART-STRATEGY-DCB-2025
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
Keywords: Complex Coronary Bifurcation; Upfront 2-stenting; Upfront Drug-coated Balloon; Side Branch; Prognosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, open-label, randomized controlled, superiority trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical outcome assessment will be performed under blinded assessment about the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upfront DCB-based hybrid strategy (Experimental): In upfront DCB-based hybrid strategy group, stepwise provisional strategy with side branch DCB angioplasty will be performed according to the follow standardized procedural steps. In this group, provisional stenting strategy will be performed in accordance with the European Bifurcation Club (EBC) consensus. Bail-out stenting will be performed using operator's preferred technique (e.g. T, TAP, culotte) when there will be one of the following after hybrid strategy: <TIMI 3 flow in the side branch, severe (>90%) ostial pinching, or flow-limiting dissection.
  Interventions: Other: Upfront DCB-based hybrid strategy
- Upfront 2-stenting strategy (Active Comparator): In upfront 2-stenting strategy group, systematic planned 2-stenting will be performed according to EBC recommendations. The stent technique will be at the discretion of the operator but could be one of culotte, DK-culotte, mini-crush, DK-crush, T or TAP.
  Interventions: Other: Upfront 2-stenting strategy

INTERVENTIONS:
Other: Upfront DCB-based hybrid strategy — In upfront DCB-based hybrid strategy group, stepwise provisional strategy with side branch DCB angioplasty will be performed according to the follow standardized procedural steps. In this group, provisional stenting strategy will be performed in accordance with the European Bifurcation Club (EBC) consensus. Bail-out stenting will be performed using operator's preferred technique (e.g. T, TAP, culotte) when there will be one of the following after hybrid strategy: <TIMI 3 flow in the side branch, severe (>90%) ostial pinching, or flow-limiting dissection.
  Arms: Upfront DCB-based hybrid strategy
Other: Upfront 2-stenting strategy — In upfront 2-stenting strategy group, systematic planned 2-stenting will be performed according to EBC recommendations. The stent technique will be at the discretion of the operator but could be one of culotte, DK-culotte, mini-crush, DK-crush, T or TAP.
  Arms: Upfront 2-stenting strategy

SUMMARY:
A prospective, multi-center, open-label, randomized controlled, superiority trial. The aim of the study is to compare clinical outcomes between upfront 2-stenting strategy versus upfront drug-coated balloon (DCB)-based hybrid strategy in patients with complex coronary bifurcation with clinically relevant side branch lesions.

DETAILED DESCRIPTION:
Among complex coronary artery lesions, percutaneous coronary intervention (PCI) for true bifurcation lesions has been challenging to perform and associated with a higher risk of mortality, unplanned repeat revascularization or stent thrombosis.15-17 Although current guidelines recommend 1-stenting with provisional side branch approach as an initial treatment strategy for the bifurcation lesions based on previous trials,11,12,18-22 there are studies that demonstrate better or similar outcomes with the upfront 2-stenting strategy.3,4,21,23 Of note, these trials that have favored upfront 2-stenting strategy have shown a tendency for better efficacy of 2-stenting as the severity of bifurcation lesions increases.3,4,21,23 Considering that the discrepancy among study results could be attributable to the complexity of true bifurcation lesions, it can be argued that 1-stenting with provisional SB approach by conventional balloon dilatation shows limitations in dealing with severely complex true bifurcation lesions.

During provisional stenting, unplanned side branch stenting is associated with worse clinical outcomes.24 In addition, SB failure occurred more frequently than main vessel failure in both 1-stenting and 2-stenting group.25 Considering these results, there have been some studies trying to demonstrate the effect of drug-coated balloon (DCB) angioplasty at side branch during the PCI for bifurcation lesions.5,26 In the most recent trial, DCB angioplasty yielded better results compared to conventional simple balloon dilatation.5 Thus, for true bifurcation lesions, upfront DCB-based hybrid strategy could serve as a good alternative treatment strategy that improves clinical outcomes for patients with complex coronary bifurcation lesion with clinically relevant side branch.

On this background, this trial sought to compare the clinical outcomes between upfront DCB-based hybrid strategy and upfront 2-stenting strategy in patients with complex coronary bifurcation with clinically relevant side branch.

ELIGIBILITY:
Inclusion Criteria

* Subject must be at least 19 years of age
* Patients with acute or chronic coronary syndrome intended for percutaneous coronary intervention (PCI)
* Patients with de novo complex coronary bifurcation with clinically relevant side branch. Definition of complex coronary bifurcation with clinically relevant side branch is true bifurcation lesion (Medina 1,1,1 / 1,0,1 / 0,1,1) with side branch lesion length ≥10mm and should meet at least one of the below criteria.

  i. Left main bifurcation with side branch stenosis severity ≥70% by visual estimation ii. Non-left main bifurcation with side branch reference vessel diameter ≥2.75mm and stenosis severity ≥90% by visual estimation
* Subject who can verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive approach and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria

* Hemodynamically unstable condition (SBP <90 mmHg even after administration of vasopressor, ventricular arrhythmias, or cardiogenic shock)
* Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
* Known significant congenital, severe valvular or cardiomyopathic (hypertrophic or dilated cardiomyopathy, or any other forms) process which could explain cardiac symptoms.
* Severe left ventricular systolic dysfunction (ejection fraction <30%)
* Intolerance to aspirin, clopidogrel, ticagrelor, prasugrel, or heparin.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event (MACE) | 1 year after last patient enrollment
  MACE (a composite of death, MI, clinically-driven target-vessel revascularization), according to the Academic Research Consortium (ARC) II-consensus.

SECONDARY OUTCOMES:
All-cause death | 1 year after last patient enrollment
  All-cause death
Cardiac death | 1 year after last patient enrollment
  Cardiac death
Any MI (myocardial infarction) | 1 year after last patient enrollment
  Any MI, defined by Fourth Universal definition of M
Spontaneous MI (myocardial infarction) | 1 year after last patient enrollment
  Spontaneous MI (myocardial infarction), defined by Fourth Universal definition of MI
Procedure-related MI (myocardial infarction) | 1 year after last patient enrollment
  Procedure-related MI (myocardial infarction), defined by ARC II definition
Stent thrombosis | 1 year after last patient enrollment
  Stent thrombosis, defined by ARC II definition
Unplanned revascularization (clinically-driven) | 1 year after last patient enrollment
  Unplanned revascularization (clinically-driven)
Target-vessel revascularization (clinically-driven) | 1 year after last patient enrollment
  Target-vessel revascularization (clinically-driven)
Cerebrovascular accidents (ischemic or hemorrhagic) | 1 year after last patient enrollment
  Cerebrovascular accidents (ischemic or hemorrhagic)
Bleeding (BARC 2, 3, or 5) | 1 year after last patient enrollment
  Bleeding (BARC 2, 3, or 5)
Seattle Angina Questionnaire (SAQ) (angina severity) | 1 year after last patient enrollment
  Seattle Angina Questionnaire (SAQ) (angina severity)
Procedure-related complications during index procedure | 1 year after last patient enrollment
  Procedure-related complications during index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Young Bin Song, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After completion of primary trial report, executive committee members will have discussion about sharing the individual participant data (IPD) upon reasonable requests,
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion of primary trial report
Access Criteria: Upon reasonable requests, executive committee members will have discussion about sharing the individual participant data (IPD).